CLINICAL TRIAL: NCT05849558
Title: Multi-Center, Randomized, Control, Phase IV Trial to Compare the Efficacy & Safety of Ursoplus® Capsules (UDCA 250mg & Silymarin 140mg) Versus UDCA Alone Versus Placebo Among Compensated Chronic Liver Diseased Patients
Brief Title: Study to Compare the Efficacy & Safety of Ursoplus Capsules vs. UDCA vs. Placebo Among Chronic Liver Disease Patients
Acronym: URSO-003
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URSO - 003
Record Dates: First submitted 2023-04-12; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: Group 1: with non-cirrhosis, F0, F1 and F2 Group 2: with advanced fibrosis and cirrhosis, F3 and F4
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) (Experimental): Ursoplus® capsules: UDCA 250mg & Silymarin 140mg
  2 Capsules every 12 hours
  Interventions: Drug: Ursoplus
- UDCA 250mg (Active Comparator): UDCA capsules: UDCA 250mg
  2 Capsules every 12 hours
  Interventions: Drug: UDCA 250mg
- Placebo (Placebo Comparator): Placebo alone
  2 Capsules every 12 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ursoplus — Ursoplus® capsules (UDCA 250mg & Silymarin 140mg)
  Arms: Ursoplus® capsules (UDCA 250mg & Silymarin 140mg)
Drug: UDCA 250mg — UDCA 250mg alone
  Arms: UDCA 250mg
Other: Placebo — Placebo alone
  Arms: Placebo

SUMMARY:
This study aims to compare the efficacy & safety of Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) versus UDCA alone versus Placebo among Compensated Chronic Liver Diseased Patients

DETAILED DESCRIPTION:
Research Question:

Compare the efficacy & safety of Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) versus UDCA alone versus Placebo among Compensated chronic liver diseased patients

Primary Objective:

To assess the efficacy of Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) versus UDCA 250mg alone and versus Placebo in the reduction of total serum bilirubin, Direct serum bilirubin and elevated liver Enzymes from baseline to End of Treatment (EOT)

Secondary Objectives:

* To assess the efficacy of Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) versus UDCA 250 mg alone and versus Placebo in reducing the degree of steatosis as measured by Vibration-controlled transient elastography with Controlled Attenuation Parameter (CAP)
* To assess the safety of Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) versus UDCA 250 mg alone and versus Placebo among compensated Chronic Liver Diseased Patients
* To describe improvement in quality of life for patients after treatment

A study population of 297 patients suffering from compensated chronic Liver Disease, who will be randomized according to Vibration-controlled transient elastography in screening visit into 2 groups:

* Group 1: with non-cirrhosis, F0, F1 and F2.
* Group 2: with advanced fibrosis and cirrhosis, F3 and F4.

Each group will receive either Ursoplus® capsules (UDCA 250mg & Silymarin 140mg), or UDCA alone or Placebo, through Stratified random sampling.

Duration for enrollment: 6 months Total duration of the study/subject will be approximately: 6 months for treatment and follow-up visits including the screening visit

Subjects will be enrolled for a duration of 6 months including the screening visit

* Screening visit 1 (Treatment initiation)
* Visit 2: after 1st month, follow-up 1
* Visit 3: after 2nd month, follow-up 2
* Visit 4: after 3rd month, follow-up 3
* Visit 5: after 4th month, follow-up 4
* Visit 6: after 5th month, follow-up 5
* End of Study visit, after 6th month of treatment, follow-up 6

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18
2. Subjects with Compensated Chronic Liver Disease, defined as child 5-7.
3. Patients with mild disturbance of liver biochemical profile (elevated Total Serum Bilirubin ≤ 3 mg/dl, or elevated Direct Serum Bilirubin ≤ 2 mg/dl, or elevated one or more of liver enzymes, up to 3 times of the normal level (Alanine Transaminase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) & Gamma Glutamyl Transpeptidase (GGT)).
4. Non-diabetic subjects and subjects with Controlled DM-type 1 and 2 patients, HbA1C up to 7.5%
5. Non-pregnant or lactating female patients
6. Subjects who are willing to sign Informed Consent Form (ICF) and ready to comply with the protocol for the duration of the study

Exclusion Criteria:

1. Subjects with a history of hypersensitivity to any of the ingredients of the medications being studied
2. Subjects with positive PCR/or antibodies to Hepatitis C in the past 6 months
3. Subjects with positive hepatitis B surface antigen (HBsAg)
4. Subjects with elevated liver enzymes more than 3 times of the normal level Alanine Transaminase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) & Gamma Glutamyl Transpeptidase (GGT).
5. Subjects with Primary Biliary Cirrhosis (PBC) and Primary Sclerosing Cholangitis (PSC).
6. Subjects with Child Pugh Score more than 7.
7. Subjects with history of bleeding varices.
8. Subjects having uncontrolled Diabetes (HbA1cmore than 7.5 %)
9. Subjects with any medical condition requiring the usage of medication that may interfere with the absorption, distribution, metabolism or excretion of the study drug such as:

   1. Bile acid sequestering agents such as cholestyramine and colestipol.
   2. Antacids containing aluminum hydroxide.
   3. Drugs affecting lipid metabolism such as estrogens, oral and hormonal contraceptives, and clofibrate (and perhaps other lipid-lowering drugs)
10. Subjects who are receiving other liver support drugs (including drugs of the study), 1 month before study initiation.
11. Subjects with auto immune liver disease taking corticosteroid or immune suppressant
12. Pregnant or breast-feeding women
13. Use of oral contraceptives in child bearing ladies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Total serum bilirubin | Up to 6 months
  Change in mean Total serum bilirubin from baseline (visit 1) to End of study between the 3 treatment groups
Change in Direct Serum Bilirubin | Up to 6 months
  Change in mean Direct Serum Bilirubin from baseline (visit 1) to End of study between the 3 treatment groups
Change in Elevated Liver Enzymes | Up to 6 months
  Change in mean AST & ALT from baseline (visit 1) to End of study between the 3 treatment groups

SECONDARY OUTCOMES:
Improved degree of Steatosis | Up to 6 months
  Change in the mean score of Controlled Attenuation Parameter (CAP) from baseline (visit 1) to End of study between the 3 treatment groups, measured by Vibration-controlled transient elastography
Improved quality of life | Up to 6 months
  Change in the mean Score of different items of the RAND 36-Item Health Survey between the 3 treatment groups after 3 months (visit 4) and 6 months of treatment (End of study visit).
Incidence of adverse events (AEs) | Up to 6 months
  Percent of serious (SAEs)/ non-serious adverse events (AEs), including percent changes in lab tests and percent of AEs leading to permanent discontinuation of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Dr Esmat, PhD, Principal Investigator — Air Force Specialized Hospital; Mohamed El Kassas, PhD, Principal Investigator — Helwan University Hospital
Locations (1):
- Air Force Specialized Hospital, Cairo, New Cairo, Egypt

DOCUMENTS (4):
  • Study Protocol (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05849558/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05849558/SAP_001.pdf
  • Informed Consent Form: AFSH Hospital (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05849558/ICF_002.pdf
  • Informed Consent Form: Helwan University (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05849558/ICF_003.pdf